CLINICAL TRIAL: NCT00977717
Title: Pharmacogenomic Study to Predict Toxicity and Response in Colorectal Cancer Patients Treated With Oxaliplatin-based Chemotherapy
Brief Title: Pharmacogenomic Study to Predict Neurotoxicity of Oxaliplatin
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Se Hoon Park, MD, Samsung Medical Center, Seoul, Korea
Other Study IDs: 2008-05-052
Record Dates: First submitted 2009-09-03; First posted 2009-09-16 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2010-04

CONDITIONS: Curatively Resected Stage III Colon Cancer
Keywords: oxaliplatin; neuropathy; SNPs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from peripheral blood samples using DNA isolation kit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FOLFOX: Stage III colorectal cancer patients who are treated with adjuvant FOLFOX chemotherapy

SUMMARY:
In order to explore genetic factors that may determine the neurotoxicity of oxaliplatin-based chemotherapy, germinal gene polymorphisms will be analyzed.

DETAILED DESCRIPTION:
To investigate the impact of single nucleotide (SNP) polymorphism on the toxicity profile in colorectal cancer patients treated with FOLFOX chemotherapy, 10 cc of blood will be drawn in EDTA tube for extraction. DNA will be extracted from peripheral blood samples using DNA isolation kit, and SNP polymorphisms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* curatively resected colon adenocarcinoma
* pathologically staged III
* adequate performance status
* adequate major organ functions
* to be treated with adjuvant FOLFOX chemotherapy
* written informed consent

Exclusion Criteria:

* those who disagree the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Curatively resected stage III colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
neuropathy | six months

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Baek KK, Lee J, Park SH, Park JO, Park YS, Lim HY, Kang WK, Cho YB, Yun SH, Kim HC, Lee WY, Chun HK. Oxaliplatin-induced chronic peripheral neurotoxicity: a prospective analysis in patients with colorectal cancer. Cancer Res Treat. 2010 Dec;42(4):185-90. doi: 10.4143/crt.2010.42.4.185. Epub 2010 Dec 31. PMID 21253319